CLINICAL TRIAL: NCT02933892
Title: Benefit of Transradial Approach in Chronic Kidney Disease Population Undergoing Cardiac Catheterization, A Single Center Randomized Controlled Trial
Brief Title: Benefit of Transradial Approach in Chronic Kidney Disease Population Undergoing Cardiac Catheterization
Acronym: RADIAL-CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L16-092
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease; Acute Kidney Injury; Heart Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Heart Diseases | interventions — Cardiac Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transradial Access (Active Comparator): Patients scheduled for cardiac catheterization will be randomly assigned to have the doctor insert the catheter via the arm access site (transradial access).
  Interventions: Procedure: Cardiac Catheterization
- Transfemoral Access (Active Comparator): Patients scheduled for cardiac catheterization will be randomly assigned to have the doctor insert the catheter via the inner thigh access site (transfemoral access).
  Interventions: Procedure: Cardiac Catheterization

INTERVENTIONS:
Procedure: Cardiac Catheterization — Cardiac catheterization is a diagnostic procedure used to treat and diagnose heart conditions.

SUMMARY:
The investigators will conduct a randomized controlled trial that aims to compare the incidence of contrast-induced nephropathy between transradial- and transfemoral-access cardiac catheterization.

DETAILED DESCRIPTION:
Cardiac catheterization is a medical procedure used to diagnose and treat heart conditions. Approaching the heart can be done by different access sites: via the femoral artery (transfemoral) or the radial artery (transradial). Transfemoral access (TFA) is the primary mode of arterial access. Several clinical trials have demonstrated the benefit of transradial over transfemoral approach. The primary advantage of transradial approach is a significant reduction of access-site complications. Chronic Kidney Disease (CKD) is a serious condition associated with premature mortality, decreased quality of life, and increased health-care expenditures. ). It is commonly found in patients with diabetes, hypertension, hyperlipidemia, coronary artery disease, or combinations of these risk factors. Coronary artery disease and CKD are often comorbid conditions seen in the cath lab. Cardiac catheterization is a mainstay of diagnosis and treatment for coronary artery disease and 58% of deaths in CKD are related to cardiovascular deaths. Patients with CKD and who undergo a cardiac catheterization are at risk for contrast-induced nephropathy (CIN) due to the dye used during the procedure.

The investigators will conduct a randomized controlled trial that aims to compare the incidence of CIN between transradial and transfemoral cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo non-emergent cardiac catheterization at University Medical Center Hospital, Lubbock, TX from January 2016 to January 2018. Emergent cardiac catheterizations will be defined as a catheterization scheduled < 24 hours from a cardiac event.
2. Patients willing to be randomized to TFA or TRA procedure.
3. Patients signed and dated the informed consent agreeing to participate in the study.
4. Patients with chronic kidney disease, defined as eGFR = 15-59mL/min defined by the MDRD formula. (eGFR is a standard of care measurement for all patients undergoing coronary intervention.).
5. Patients ages 18-88 years old.

Exclusion Criteria:

1. Patients who have previously undergone a coronary artery bypass graft procedure.
2. Patients with prior catheterization within the last 5 years.
3. Women who are pregnant or expect to become pregnant. Pregnancy tests for women of childbearing potential (WOCHP) will be performed as standard of care.
4. Patients with a history of cardiogenic shock.
5. Children (under the age of 18).
6. Medical, geographical, or social factors making study participation impractical, i.e. documented noncompliance, unable to return for follow-ups and lab draws, etc.
7. A positive Allen's Test on the right radial artery.
8. Any condition preventing TRA or TFA access.
9. Contrast used within the previous 3 weeks.
10. Allergy to contrast dye.
11. Inability to successfully access the artery randomized to use.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10; Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of CIN | 3 days
Incidence of CIN | 30 days
Need for dialysis | 30 days

SECONDARY OUTCOMES:
All cause mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Subasit Acharji, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, the research group may be potentially interested in sending data for further analyses.

REFERENCES:
- [Background] Caputo RP, Tremmel JA, Rao S, Gilchrist IC, Pyne C, Pancholy S, Frasier D, Gulati R, Skelding K, Bertrand O, Patel T. Transradial arterial access for coronary and peripheral procedures: executive summary by the Transradial Committee of the SCAI. Catheter Cardiovasc Interv. 2011 Nov 15;78(6):823-39. doi: 10.1002/ccd.23052. Epub 2011 May 4. PMID 21544927
- [Background] Bertrand OF, Belisle P, Joyal D, Costerousse O, Rao SV, Jolly SS, Meerkin D, Joseph L. Comparison of transradial and femoral approaches for percutaneous coronary interventions: a systematic review and hierarchical Bayesian meta-analysis. Am Heart J. 2012 Apr;163(4):632-48. doi: 10.1016/j.ahj.2012.01.015. PMID 22520530
- [Background] Vassalotti JA, Centor R, Turner BJ, Greer RC, Choi M, Sequist TD; National Kidney Foundation Kidney Disease Outcomes Quality Initiative. Practical Approach to Detection and Management of Chronic Kidney Disease for the Primary Care Clinician. Am J Med. 2016 Feb;129(2):153-162.e7. doi: 10.1016/j.amjmed.2015.08.025. Epub 2015 Sep 25. PMID 26391748
- [Background] Tonelli M, Wiebe N, Culleton B, House A, Rabbat C, Fok M, McAlister F, Garg AX. Chronic kidney disease and mortality risk: a systematic review. J Am Soc Nephrol. 2006 Jul;17(7):2034-47. doi: 10.1681/ASN.2005101085. Epub 2006 May 31. PMID 16738019
- [Background] Parfrey PS, Griffiths SM, Barrett BJ, Paul MD, Genge M, Withers J, Farid N, McManamon PJ. Contrast material-induced renal failure in patients with diabetes mellitus, renal insufficiency, or both. A prospective controlled study. N Engl J Med. 1989 Jan 19;320(3):143-9. doi: 10.1056/NEJM198901193200303. PMID 2643041
- [Background] Haase M, Bellomo R, Matalanis G, Calzavacca P, Dragun D, Haase-Fielitz A. A comparison of the RIFLE and Acute Kidney Injury Network classifications for cardiac surgery-associated acute kidney injury: a prospective cohort study. J Thorac Cardiovasc Surg. 2009 Dec;138(6):1370-6. doi: 10.1016/j.jtcvs.2009.07.007. Epub 2009 Sep 5. PMID 19733864
- [Background] Dangas G, Iakovou I, Nikolsky E, Aymong ED, Mintz GS, Kipshidze NN, Lansky AJ, Moussa I, Stone GW, Moses JW, Leon MB, Mehran R. Contrast-induced nephropathy after percutaneous coronary interventions in relation to chronic kidney disease and hemodynamic variables. Am J Cardiol. 2005 Jan 1;95(1):13-9. doi: 10.1016/j.amjcard.2004.08.056. PMID 15619387
- [Background] Ohno Y, Maekawa Y, Miyata H, Inoue S, Ishikawa S, Sueyoshi K, Noma S, Kawamura A, Kohsaka S, Fukuda K. Impact of periprocedural bleeding on incidence of contrast-induced acute kidney injury in patients treated with percutaneous coronary intervention. J Am Coll Cardiol. 2013 Oct 1;62(14):1260-1266. doi: 10.1016/j.jacc.2013.03.086. Epub 2013 Jun 12. PMID 23770181
- [Background] Vuurmans T, Byrne J, Fretz E, Janssen C, Hilton JD, Klinke WP, Djurdjev O, Levin A. Chronic kidney injury in patients after cardiac catheterisation or percutaneous coronary intervention: a comparison of radial and femoral approaches (from the British Columbia Cardiac and Renal Registries). Heart. 2010 Oct;96(19):1538-42. doi: 10.1136/hrt.2009.192294. Epub 2010 Jul 28. PMID 20668106
- [Background] Kooiman J, Seth M, Dixon S, Wohns D, LaLonde T, Rao SV, Gurm HS. Risk of acute kidney injury after percutaneous coronary interventions using radial versus femoral vascular access: insights from the Blue Cross Blue Shield of Michigan Cardiovascular Consortium. Circ Cardiovasc Interv. 2014 Apr;7(2):190-8. doi: 10.1161/CIRCINTERVENTIONS.113.000778. Epub 2014 Feb 25. PMID 24569598
- [Background] Sunder S, Jayaraman R, Mahapatra HS, Sathi S, Ramanan V, Kanchi P, Gupta A, Daksh SK, Ram P. Estimation of renal function in the intensive care unit: the covert concepts brought to light. J Intensive Care. 2014 May 7;2(1):31. doi: 10.1186/2052-0492-2-31. eCollection 2014. PMID 25520843
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671